CLINICAL TRIAL: NCT06728332
Title: ESTeeM: Evaluation of Sleep Disturbances in Menopause
Brief Title: An Observational Study to Learn More About How Menopause Affects Women's Sleep and How They Are Being Treated for Sleep Problems
Acronym: ESTeeM
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 22815
Record Dates: First submitted 2024-11-13; First posted 2024-12-11 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Sleep Disturbances Associated With Menopause

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: Females experiencing sleep disturbances associated with menopause
  Interventions: Other: No study intervention

INTERVENTIONS:
Other: No study intervention — No visits or examinations, laboratory tests or procedures are mandated or required for this study. Providers in the study recruitment network will recruit eligible patients through an existing visit. After this referral, the study is conducted entirely electronically.

SUMMARY:
This is an observational study in which data from women with sleep disturbances and vasomotor symptoms, also known as hot flashes, associated with menopause (SDM) are collected and studied.

Menopause is part of a natural aging process and happens when women's menstrual cycles, also called periods, stop. Sleep disturbances, such as frequent waking up at night, are a common symptom (clinical sign) and a major worry associated with menopause that affects women's quality of life.

The participants will continue to take their regular treatment for their SDM as agreed with their doctors. These are called "standard of care" treatments.

Because both patients and doctors don't know much about SDM, women are often treated with sleep medicines that can lead to addiction and cause side effects. This study will help us to learn more about how much menopause-related sleep problems affect a woman's overall health and well-being. We also want to find out how women are currently being treated or treat themselves for these sleep problems, so we can figure out if there's a need for new treatments that focus specifically on menopause-related sleep issues

To do this, researchers will collect information on:

* the number of times a woman wakes up during the night and the total time she is awake after she first falls asleep
* the time when a woman goes to bed and when she wakes up in the morning
* how long it takes for a woman to fall asleep after going to bed
* changes in sleep problem questionnaire scores to assess how these problems affect a woman's quality of life

The data will come from combining all the electronic health record databases, patient related questionnaires, and data from smartwatches that the women will wear on their wrists. The data will be collected between November 2024 to May 2025.

In this study, researchers will combine all the electronic data during a 28-day follow-up period. No visits or tests are required as part of this study.

ELIGIBILITY:
Inclusion Criteria:

* Women experiencing menopause assigned female at birth, 40-65 years of age, residing in the United States.

  o Where being in the menopausal period is defined as at least 12 months of spontaneous amenorrhea prior to index date (the date informed consent was signed) or surgical bilateral oophorectomy with or without hysterectomy at least 6 weeks prior to index date.
* Sleep disturbances due to menopause, defined as self-reported disturbances characterized by waking up at night and/or poor quality of sleep (including difficulty falling asleep, short sleep, waking up early).
* Signed ICF by the patient.
* Provided access to medical records, directly granting access through the HRS platform and the provider's portal or providing contact information and a medical records release form.

Exclusion Criteria:

* Menopause induced chemically or from radiation therapy (i.e., chemotherapy).
* Medical conditions that impact sleep, including diagnosed chronic insomnia, sleep apnea, restless leg syndrome, circadian rhythm sleep disorder; current or history (except complete remission for 5 years or more) of any malignancy (except basal and squamous cell skin tumors).
* Women self-reporting being under the care of a HCP for suicidal ideation in the past six months, clinical anxiety in the past six months, or clinical depression in the past six months.
* Patients participating in a clinical trial.
* Pregnant women.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Women experiencing menopause assigned female at birth
Study Population: Females from 40 to 65 years (inclusive) experiencing sleep disturbances associated with menopause.
Sampling Method: Non-Probability Sample
Enrollment: 750 (Actual)
Dates: Start 2024-12-06 (Actual); Primary Completion 2025-08-29 (Actual); Study Completion 2025-10-27 (Actual)

PRIMARY OUTCOMES:
Number of awakenings in the night. | From Day 1 to Day 28.
Mean WASO (wakefulness after sleep onset) | From Day 1 to Day 28
  Total number of minutes that a participant is awake after having initially fallen asleep
Mean number of moderate or severe hot flashes per night | From Day 1 to Day 28
Mean sleep efficiency score | From Day 1 to Day 28
  Defined as the percentage of time spent asleep while in bed
Mean length of time (in minutes) to fall asleep | From Day 1 to Day 28
Mean total sleep disturbance score (T-score) derived from PROMIS-SD-SF-8b | Day 1, Day 14 and Day 28
  PROMIS-SD-SF-8B: Patient-reported Outcomes Measurement Information System Sleep disturbance short form 8b.
Menopause-specific quality-of-life questionnaire (MENQOL) total score | Day 1, Day 14 and Day 28
  Measured by ePRO.
Insomnia Severity Index (ISI) total Score | Day 1, Day 14 and Day 28
Socioeconomic status short-form questionnaire | Day 0

SECONDARY OUTCOMES:
Descriptive analysis of demographics | Day 0
Descriptive analysis of clinical characteristics | Day 0
Lifestyle questionnaire | Day 0
  Questionnaire includes smoking history, alcohol consumption, caffeine consumption, other persons in the home and work schedule.
Comorbid conditions and dates of diagnosis from patient EHR (electronic health record) | Day 0
Concomitant medications, from patient medication survey | Day 0
Body mass index (BMI) | Day 0
Number of previous pregnancies from patient EHR | Day 0
Non-pharmacologic treatments for sleep disturbances | Day 0
Number of EHR (electronic Health record) documented prescriptions for sleep disturbances. | Retrospective analysis from 12 months prior to ICF
Number of patient-reported medications and supplements for sleep disturbances. | From 6 months prior Day 1
Number of patients reporting alternative treatment/management for sleep disturbances | Day 0
Questionnaire of satisfaction score for medications and supplements used to treat sleep disturbances. | From 6 months prior Day 1
Names of prescription and non-prescription medications and supplements for sleep disturbances reported in Daily Morning Diaries, including dosage. | Day 1 to Day 28
List of types of treatment formerly prescribed for sleep disturbances, from patient medication survey. | Day 0
Duration of treatments formerly prescribed for sleep disturbances, by drug class, from patient medication survey. | Day 0
Proportion of days PRN medication used. | From Day 1 to Day 28
Among medications for sleep disturbances discontinued within 6 months of enrollment, patient reported reason for discontinuation. | Day 0
HADS (Hospital Anxiety and Depression Scale) total score. | Day 0

CONTACTS AND LOCATIONS:
Locations (1):
- Bayer, Whippany, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.